CLINICAL TRIAL: NCT02051556
Title: Working on Asymmetry in Parkinson's Disease: a Double Blind, Randomized, Controlled Rehabilitation Trial.
Brief Title: Working on Asymmetry in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Nicola Modugno, MD, PhD, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ASPD-01
Record Dates: First submitted 2014-01-16; First posted 2014-01-31 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Freezing of gait; Asymmetry; Rehabilitation; Physical therapy
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Best Side Improvement (Experimental): Physical Therapy BSI (Best Side Improvement), aimed to potentiate the less affected body side.
  Interventions: Behavioral: Physical Therapy BSI
- Worse side improvement (Experimental): Physical Therapy WSI (Worst Side Improvement), aimed to potentiate the most affected body side.
  Interventions: Behavioral: Physical Therapy WSI
- Standard treatment (Active Comparator): Physical Therapy ST (Standard Treatment), aimed to potentiate both sides equally.
  Interventions: Behavioral: Physical Therapy ST

INTERVENTIONS:
Behavioral: Physical Therapy WSI — Each session has duration of one hour and includes a first part of warming up, a final part of cooling down (these two parts were the same for all the groups) and an active part that includes exercises with a number of repetitions according to the aim of potentiating the most affected side (WSI).
  Arms: Worse side improvement
Behavioral: Physical Therapy BSI — Each session has duration of one hour and includes a first part of warming up, a final part of cooling down (these two parts were the same for all the groups) and an active part that includes exercises with a number of repetitions according to the aim of potentiating the least affected side (BSI).
  Arms: Best Side Improvement
Behavioral: Physical Therapy ST — Each session has duration of one hour and includes a first part of warming up, a final part of cooling down and an active part that includes exercises with a number of repetitions according to the aim of potentiating both sides equally (ST). In this case the number of repetitions was the same for both sides.
  Arms: Standard treatment

SUMMARY:
Freezing of gait (FOG) is a disabling episodic gait disturbance that is common among patients with Parkinson's disease (PD). The symptoms of PD generally show an asymmetric onset and progression.

In particular, impairments in rhythmicity, symmetry, and bilateral coordination have been reported to be associated with FOG episodes. As the maintenance of gait depends on the precise alternating movements of both legs, irregularities in rhythm, symmetry, and bilateral coordination may impair gait sequence, potentially causing freezing.

Results of recent studies strongly suggest that bilateral uncoordinated gait and marked gait asymmetry are associated with FOG. Moreover, it has recently been hypothesized that this may lead to a degree of asymmetric motor function, and that FOG in parkinsonian patients is triggered by a breakdown in the bilateral co-ordination underlying the normal timing of gait. Aim of the study was to evaluate how the modulation of asymmetry through physical therapy might improve gait and FOG.

DETAILED DESCRIPTION:
The patients will be'blind' to the study protocol and will be randomly assigned to one of the three study arms: 1) physiotherapy aimed to potentiate the more affected body side (worst side improvement, WSI); 2) physiotherapy aimed to potentiate the less affected body side (best side improvement, BSI); 3) physiotherapy aimed to potentiate both sides equally (standard treatment, ST). Each group will be undergo physiotherapy twice a week for three months. Each session will have duration of one hour and include a first part of warming up, a final part of cooling down (these two parts are the same for all the groups) and an active part (which is different from group to group). The active part includes exercises which are alike for all the groups but with a number of repetitions different from group to group according to the aim of potentiating the most affected side (WSI) or the least affected side (BSI) or both sides equally (in this case the number of repetitions was the same for both sides; ST). Medical treatment will be kept stable through all the study duration; medications are expressed as levodopa daily dose equivalent (LEDD).

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease, freezing of gait history, informed consent

Exclusion Criteria:

* depression, severe orthopedic diseases

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Motor Symptoms | 24 weeks

SECONDARY OUTCOMES:
Freezing of gait | 24 weeks

OTHER OUTCOMES:
Short physical performance battery | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Modugno, MD, PhD, Study Chair — IRCCS NEUROMED
Locations (1):
- Irccs Neuromed, Pozzilli, Isernia, Italy

REFERENCES:
- [Result] Modugno N, Iaconelli S, Fiorlli M, Lena F, Kusch I, Mirabella G. Active theater as a complementary therapy for Parkinson's disease rehabilitation: a pilot study. ScientificWorldJournal. 2010 Nov 16;10:2301-13. doi: 10.1100/tsw.2010.221. PMID 21103799